CLINICAL TRIAL: NCT04373889
Title: SARS-COV-2 Prevalence, Seroprevalence and Seroconversion Among Healthcare Workers in Belgium During the 2020 COVID-19 Outbreak
Brief Title: COVID-19 Among Healthcare Workers in Belgian Hospitals
Acronym: COVHECBEHO
Status: Completed | Type: Observational
Sponsor: Sciensano (Other Government)
Collaborators: Institute of Tropical Medicine, Belgium (Other)
Responsible Party: Sponsor
Other Study IDs: Sciensano
Record Dates: First submitted 2020-04-13; First posted 2020-05-05 (Actual); Last update posted 2021-10-04 (Actual); Status verified 2021-10

CONDITIONS: SARS-CoV-2; COVID-19
Keywords: SARS-CoV-2; COVID-19; Hospital healthcare workers; Belgium; Pandemic 2020; Hospital
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Due to the situation this study, originally planted until September 2020, was extended with 7 months until April 2021. This extension was approved by the ethical committee University hospital Ghent, Belgium.

The novel SARS-CoV-2 (Severe Acute Respiratory Syndrome-associated Coronavirus type 2) is rapidly spreading over the world causing a condition called Coronavirus disease 2019 (COVID-19). Hospital health care workers (HCW) have received detailed instructions to protect themselves against this infection, but it is likely that at least some of the HCW will get infected either at their workplace or elsewhere. It would be useful to document prevalence and seroprevalence of SARS-CoV-2 and their monthly evolution among Belgian active hospital HCW during a period of 12 months starting beginning of April 2020 and the number of new cases (incidence) of COVID-19 and SARS-CoV-2 seroconversions among Belgian hospital HCW during a period of 12 months which are the primary objectives of this study.

Additionally the study will validate serological tests (subject to change/addition depending on the evolution of scientific research) against the plaque reduction neutralization test (PRNT) (gold standard); validate the saliva sample (sampling with Oracol or equivalent) against the standard naso/oro pharyngeal swabbing (NOPS) to perform RT-qPCR for SARS-CoV-2 diagnostic purposes, as well as against the standard serology (serum); validate the nasal swab against the standard (NOPS) to perform RT-qPCR for SARS-CoV-2 for diagnostic purposes; investigate potential risk factors for the infection; quantify the proportion of asymptomatic cases among new cases that develop during a period of 12 months.

To reach these primary and secondary objectives the researchers will conduct a prospective cohort study in which a random selection of HCW currently working in Belgian hospitals will be tested monthly (with for the first month an additional testing point at 14 days). The testing will include four kind of laboratory tests, being; a molecular (PCR) test on a nasopharyngeal, a saliva and nasal sample (for nasal and saliva sample only testing until 50 PCR positive and 50 PCR negative samples are collected) and a serological test for which a blood sample is needed. To asses risk factors, at each testing point a questionnaire providing basic socio-demographic and health characteristics of the HCW including presence of symptoms since the previous testing point and the HCW's involvement in caring for COVID-19 patients will be completed.

Laboratory data and epidemiological data (questionnaire) will be collected simultaneously. In each of the participating hospitals, one contact person will be designated to coordinate the study locally (ideally a staff member of the local infection and prevention control team) and communicate with the researchers. The sample size calculation indicated the inclusion of 17 randomly selected Belgian hospitals and in each hospital 50 randomly selected HCW. HCW can only be enrolled in the study after give a written informed consent.

Laboratory testing will be performed at the Virology Diseases and Immune Response services of Sciensano, Ukkel, and the Virology Laboratory of the Institute of Tropical Medicine, Antwerp. The laboratory test results will be communicated by the laboratory to each participant. Each participant and sample will have a unique code assigned. Data collected through the questionnaire will be send psuedonymised (using the unique code) to the epidemiologist at Sciensano. The laboratory will prepare a list of test results by unique code to be linked for further analysis with the questionnaire data. None of the researchers who will analyse the data will be involved in data collection, nor in the care of COVID-19 patients.

This study is a Belgian multicentric study executed by Sciensano, Brussels, in collaboration with the Institute of Tropical Medicine, Antwerp.

ELIGIBILITY:
Inclusion Criteria:

* Any permanent medical and paramedical staff working in the hospital who provided a signed informed consent to participate in the study.
* Participants must have a social security insurance (mandatory in Belgium).
* This study only include adults.

Exclusion Criteria:

* Staff hired on a temporary (interim) basis will be excluded as follow-up over time will be compromised.
* Administrative staff or technical staff will also be excluded.
* HCW who were not active during the inclusion period will automatically be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Study population include health care workers currently working in Belgian hospitals.
  According to current national guidelines, HCW in contact with persons at risk for COVID-19 experiencing mild respiratory symptoms without fever are allowed to work if clinical condition permits, while wearing a mask and observing usual hygiene measures. Healthcare workers experiencing respiratory symptoms and fever are systematically tested and if positive, isolated at home, if negative, eventually working wearing a mask if the clinical state allows it. Those who recovered from a documented infection are also allowed to work. HCW who are not in contact with persons at risk for COVID-19 are not tested and systematically isolated in case of any unusual respiratory symptom. This implies that at baseline, the study population will only include asymptomatic or paucisymptomatic HCW applying proper infection prevention measures.
Sampling Method: Probability Sample
Enrollment: 850 (Actual)
Dates: Start 2020-04-22 (Actual); Primary Completion 2021-04-30 (Actual); Study Completion 2021-04-30 (Actual)

PRIMARY OUTCOMES:
Change of prevalence of COVID-19 infection among Belgian active hospital healthcare workers (HCW) | "Day 1", "Week 2", "Week 4", "Month 2", "Month 3", "Month 4", "Month 5", "Month 6", "Month 7", "Month 8", "Month 9", "Month 10", "Month 11" and "Month 12"
  Change in the percentage of HCW with positive RT-qPCR test on nasopharyngeal swabs among all HCW tested
Change of prevalence of COVID-19 infection among Belgian active hospital healthcare workers (HCW) | "Day 1", "Week 2", "Week 4", "Month 2", "Month 3", "Month 4", "Month 5", "Month 6", "Month 7", "Month 8", "Month 9", "Month 10", "Month 11" and "Month 12"
  Change in the absolute number of HCW with positive RT-qPCR test on nasopharyngeal swabs among the total number of all HCW tested
Change of seroprevalence of SARS-CoV-2 among Belgian active hospital HCW | "Day 1", "Week 2", "Week 4", "Month 2", "Month 3", "Month 4", "Month 5", "Month 6", "Month 7", "Month 8", "Month 9", "Month 10", "Month 11" and "Month 12"
  Change in percentage of HCW with specific SARS-CoV-2 IgG/IgM detected in their serum by ELISA (positive SARS-CoV-2 serological test) among all HCW tested
Change of seroprevalence of SARS-CoV-2 among Belgian active hospital HCW | "Day 1", "Week 2", "Week 4", "Month 2", "Month 3", "Month 4", "Month 5", "Month 6", "Month 7", "Month 8", "Month 9", "Month 10", "Month 11" and "Month 12"
  Change in the absolute number of HCW with specific SARS-CoV-2 IgG/IgM detected in their serum by ELISA (positive SARS-CoV-2 serological test) among the total number of all HCW tested
Change in new cases (incidence) of COVID-19 among Belgian hospital HCW | "Week 2", "Week 4", "Month 2", "Month 3", "Month 4", "Month 5", "Month 6", "Month 7", "Month 8", "Month 9", "Month 10", "Month 11" and "Month 12"
  Change in the percentage of HCW with positive RT-qPCR test on nasopharyngeal swabs among all HCW tested detected at each of the study follow-up testing points that did not have a positive RT-qPCR test before.
Change in new cases (incidence) of COVID-19 among Belgian hospital HCW | "Week 2", "Week 4", "Month 2", "Month 3", "Month 4", "Month 5", "Month 6", "Month 7", "Month 8", "Month 9", "Month 10", "Month 11" and "Month 12"
  Change in absolute number of HCW with positive RT-qPCR test on nasopharyngeal swabs among the total number of HCW tested detected at each of the study follow-up testing points that did not have a positive RT-qPCR test before.
Change in SARS-CoV-2 seroconversion among Belgian hospital HCW | "Week 2", "Week 4", "Month 2", "Month 3", "Month 4", "Month 5", "Month 6", "Month 7", "Month 8", "Month 9", "Month 10", "Month 11" and "Month 12"
  Change in the percentage of HCW with specific SARS-CoV-2 IgG/IgM detected in their serum by ELISA (positive SARS-CoV-2 serological test) among all HCW tested at each of the study follow-up testing points that did not have a positive SARS-CoV-2 serological test before.
Change in SARS-CoV-2 seroconversion among Belgian hospital HCW | "Week 2", "Week 4", "Month 2", "Month 3", "Month 4", "Month 5", "Month 6", "Month 7", "Month 8", "Month 9", "Month 10", "Month 11" and "Month 12"
  Change in the absolute number of HCW with specific SARS-CoV-2 IgG/IgM detected in their serum by ELISA (positive SARS-CoV-2 serological test) among the total number of HCW tested at each of the study follow-up testing points that did not have a positive SARS-CoV-2 serological test before.

SECONDARY OUTCOMES:
Sensitivity and specificity of serological tests | "Month 3"
  For serological analyses, the "background" serological positivity of the HCW to various CoV will be tested in order to have a clear view on true seroconversions. Antibody titers (IgM/IgG) against SARS-CoV-2; HKU-1 and OC-43 as well as 229-E and NL-63 will be determined in order to assess specificity and document potential seroconversion. Furthermore, the presently available serological tests need to be validated and confirmed with a plaque reduction neutralization test (PRNT). To that end researchers will use a Vero cell-based in vitro virus neutralization test.
Sensitivity and specificity of saliva sampling method (sampling with Oracol or equivalent) | "Month 3"
  RT-qPCR will be done on the matching saliva sample, enabling to validate or not saliva sampling for SARS-CoV-2 detection (calculating test sensitivity and specificity). serology will equally be performed on saliva samples enabling to validate or not the saliva sampling for antibody (IgM/IgG) detection (calculate test sensitivity and specificity).
Validate the nasal swab against the standard | "Month 3"
  RT-qPCR will be done on the matching nasal swab, enabling to validate or not nasal swab for SARS-CoV-2 detection (calculating test sensitivity and specificity)
Potential risk factors for the infection | "Month 5" and "Month 12"
  Proportion (%) infected HCW by professional exposure (specific function, specialty of ward, contact with confirmed case), and by health characteristics (co-morbidities, presence of symptoms, use of medications).
The proportion of asymptomatic cases among new cases that develop during a period of 12 months | "Month 5" and "Month 12"
  Percentage of asymptomatic cases among new cases (positive RT-qPCR or serological test) that develop during a period of 5 months
The proportion of asymptomatic cases among new cases that develop during a period of 12 months | "Month 5" and "Month 12"
  Absolute number of asymptomatic cases among new cases (positive RT-qPCR or serological test) that develop during a period of 5 months

CONTACTS AND LOCATIONS:
Locations (1):
- Sciensano, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mortgat L, Verdonck K, Hutse V, Thomas I, Barbezange C, Heyndrickx L, Fischer N, Vuylsteke B, Kabouche I, Arien KK, Desombere I, Duysburgh E. Prevalence and incidence of anti-SARS-CoV-2 antibodies among healthcare workers in Belgian hospitals before vaccination: a prospective cohort study. BMJ Open. 2021 Jun 29;11(6):e050824. doi: 10.1136/bmjopen-2021-050824. PMID 34187832